CLINICAL TRIAL: NCT03023280
Title: Radiofrequency Ablation in Patients With Large Cervical Heterotopic Gastric Mucosa and Globus Sensation
Status: Completed | Type: Observational
Sponsor: Dr. Ivan Kristo (Other)
Responsible Party: Sponsor-Investigator, Dr. Ivan Kristo, Dr.med.univ., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: 1723/2015
Record Dates: First submitted 2016-12-24; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Symptomatic Heterotopic Gastric Mucosa
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing radio frequency ablation: Patients undergoing radio frequency for large symptomatic heterotypic gastric mucosa
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation

SUMMARY:
Symptomatic heterotopic gastric mucosa also known as cervical inlet patch (CIP) may be present in varying shapes and causes symptoms of laryngopharyngeal reflux like globus sensations, hoarseness and chronic cough. Unfortunately, argon plasma coagulation, standard treatment of small symptomatic CIP, is limited for large heterotopic gastric mucosa due to concerns of stricture formation. Therefore, the investigators aimed to investigate the effect of radiofrequency ablation (RFA), a novel minimal-invasive ablation method, in the treatment of large symptomatic CIP.

ELIGIBILITY:
Inclusion Criteria:

* negative PPI trial, ph-metry without correlation on globus sensation, prior high-resolution manometry

Exclusion Criteria:

* not willing to participate in follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with macroscopic and histologic evidence of large (≥ 20mm diameter) heterotopic gastric mucosa.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Complete histologic eradication of heterotopic gastric mucosa | measured endoscopically throughout the study period. First time point of measurement is 3 months after first ablation. Further measurements are carried out 3 months after subsequent ablations up to a maximum number of three ablations.
  the change from gastric epithelium to squamous epithelium is monitored by histological sampling throughout the study period

SECONDARY OUTCOMES:
symptom assessment | measured at the beginning, 12 weeks after first ablation and 12 weeks after final endoscopic examination
  visual analog scale 0-10 (0=no interference, 10=maximum interference) is used for the symptom assessment of globus sensation
laryngopharyngeal reflux | at the beginning of the study period and 12 weeks after last endoscopic examination
  the Reflux Finding Index is used for assessment of laryngopharyngeal reflux
SF-12 quality of life | at the beginning of the study (before ablations) and 12 weeks after final endoscopic examination
number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | adverse events are assessed within the first week after interventions
  telephone calls
laryngopharyngeal reflux II | 1 year after first ablation
  the Reflux Finding Score is measured by using laryngofibroscopy to document potential absence of laryngopharyngeal reflux at the end of the study period

REFERENCES:
- [Derived] Kristo I, Rieder E, Paireder M, Schwameis K, Jomrich G, Dolak W, Parzefall T, Riegler M, Asari R, Schoppmann SF. Radiofrequency ablation in patients with large cervical heterotopic gastric mucosa and globus sensation: Closing the treatment gap. Dig Endosc. 2018 Mar;30(2):212-218. doi: 10.1111/den.12959. Epub 2017 Oct 3. PMID 28884487